CLINICAL TRIAL: NCT04097743
Title: Effect of Pain Catastrophizing on Prescription Opioid Craving
Brief Title: Pain Catastrophizing and Prescription Opioid Craving
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted due to inability to recruit the planned sample size within the funding period and study timeline.
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dokyoung Sophia You, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50771; 1K23DA048972 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping statement (Experimental): Daily practice of pain coping statements for 7 days
  Interventions: Behavioral: Coping Statement
- Control (No Intervention): No instruction about pain coping statement.

INTERVENTIONS:
Behavioral: Coping Statement — Daily practice of coping statement
  Arms: Coping statement

SUMMARY:
Adherence to prescription opioid and opioid tapering as indicated are critical for safe chronic opioid therapy for chronic pain, but this can be difficult for patients experiencing prescription opioid craving. Because pain catastrophizing is proposed as a possible treatment target by our and others' preliminary results, the proposed study aims to determine whether pain catastrophizing is a treatment target to reduce prescription opioid craving and to investigate whether negative affect and stress hormones are potential mediators. The findings from the current study will inform whether a psychology intervention to lower pain catastrophizing will reduce opioid craving, and whether psychological and physical distress as well as cognitive function will be potential mediators of the treatment effect.

DETAILED DESCRIPTION:
Chronic pain and opioid overdose are two critical public health problems in the US. About 25 million adults (11%) suffer from chronic daily pain and up to 8 million use opioids to manage chronic pain. Unfortunately, 46 people die daily from overdose of prescription opioids. For safe chronic opioid therapy for chronic pain, physicians monitor patients' adherence to prescription opioids, and reduce or discontinue the prescription as indicated. Yet, adherence and cessation are not easy for some patients and one reason is opioid craving, a strong desire or urge to use opioids. Our preliminary data show about 34% of patients on chronic opioid therapy report craving. Craving is strongly associated with opioid misuse and negative health outcomes. To date, we do not fully understand the underlying mechanisms of prescription opioid craving in chronic pain sufferers, and psychological treatment targets to reduce craving. Based on our pilot survey, patients endorsing craving reported greater pain catastrophizing than those endorsing no craving. Our other survey study also reported a positive link between pain catastrophizing and opioid craving in patients on chronic opioid therapy for chronic pain conditions. Although these findings propose a possibility that lowering pain catastrophizing may decrease opioid craving, cross-sectional observational studies are limited in investigating a causal association. Potentially, pain catastrophizing enhances stress-induced opioid craving because stress-induced opioid craving is a well-established phenomenon in studies of addiction, and pain catastrophizing is associated with greater pain and emotional distress in patients with chronic pain. Therefore, the proposed project seeks to determine: a) the effect of pain catastrophizing on prescription opioid craving in patients on chronic opioid therapy for chronic pain and b) psychological (negative affect) and physiological (cortisol, norepinephrine) distress and cognitive function as potential mediating variables. The proposed study will use the previously validated protocol to temporarily induce and reduce pain catastrophizing and assess changes in opioid craving, negative affect, and stress hormones before and after pain catastrophizing manipulation. Additionally, this proposed study prospectively administers the protocol to reduce pain catastrophizing by thinking about and rehearsing a coping statement daily for 7 days and monitor daily opioid craving, opioid use and misuse, and negative affect for 14 days. The current project is expected to characterize the role of pain catastrophizing in opioid craving and opioid misuse, and pain catastrophizing as a critical psychological treatment target for reducing prescription opioid craving and improving prescription adherence. Furthermore, the protocol to manipulate pain catastrophizing can facilitate future research to study causal mechanisms involved in pain catastrophizing and the protocol to rapidly stabilize pain catastrophizing can be used clinically to improve the health outcome of patients taking prescription opioid for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Chronic pain ( > 3months)
* Prescription opioid use (>3 months)

Exclusion Criteria:

* Current diagnosis of cancer
* Concurrent psychological therapy
* Other severe psychiatric conditions (schizophrenia, delusional disorder, psychotic disorder, dissociative disorder, and active suicidality)
* Any skin conditions on the hand (pain testing site)
* Non-English speaker
* No access to email or smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dokyoung S You, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Pain Relief Innovations Lab, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coping Statement | Control
Started | 44 | 49
Completed | 43 | 49
Not Completed | 1 | 0
Not completed — Non-compliance of the study instruction. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Statement | Control | Total
Number analyzed (Participants) | 44 | 49 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (13.4) | 61.6 (9.83) | 61.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 19 | 20 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 40 | 37 | 77
  White/Hispanic/Latino | 1 | 4 | 5
  African American/Black | 0 | 4 | 4
  Asian | 2 | 2 | 4
  American Indian or Alaska Native | 0 | 0 | 0
  Pacific Islander/Native Hawaiian | 0 | 0 | 0
  Prefer not to say | 0 | 2 | 2
  Other | 1 | 0 | 1
Opioid Craving [Count of Participants; unit: Participants]
  Craving | 27 | 27 | 54
  Non-craving | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: Craving
Description: Craving was assessed using a 0-100 Visual Analogue Scale (VAS), with higher scores indicating greater craving in the past 24 hours.
Time Frame: At day 7 (after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
score on a scale | 12.68 (20.06) | 18.49 (27.76)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.41, ANOVA; Mean Difference (Final Values) = 3.59, Standard Error of Mean 4.36

2. Primary Outcome: Craving
Description: as for outcome 1
Time Frame: At day 14 (7 days after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
score on a scale | 12.77 (12.84) | 21.40 (22.92)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.81, ANOVA; Mean Difference (Final Values) = -1.05, Standard Error of Mean 4.41

3. Secondary Outcome: Cortisol
Description: Salivary cortisol level was the mean of samples collected at wake-up, 30 minutes after waking, and at 9:00 PM. Higher scores indicate higher cortisol levels.
Time Frame: At day 7 (after intervention)
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
ug/dL | 0.41 (0.62) | 0.84 (3.19)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.39, ANOVA; Mean Difference (Final Values) = 0.41, Standard Error of Mean 0.47

4. Secondary Outcome: Cortisol
Description: Salivary cortisol level was the mean of samples collected at wake-up, 30 minutes after waking, and at 9:00 PM. Possible scores range 0.012-3.000 ug/dL. Higher scores indicate higher cortisol levels.
Time Frame: At day 14 (7 days after intervention)
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
ug/dL | 0.53 (1.62) | 0.35 (0.41)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.67, ANOVA; Mean Difference (Final Values) = -0.20, Standard Error of Mean 0.47

5. Secondary Outcome: Anxiety Symptoms
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 8-item short form was administered. 50 indicates the population mean with a standard deviation of 10. Possible T-Scores range from 20 - 80 and Higher scores indicate greater anxiety symptoms.
Time Frame: At day 7 (after intervention)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
T-score | 52.27 (8.88) | 50.14 (8.31)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.99, ANOVA; Mean Difference (Final Values) = 0.02, Standard Error of Mean 1.47

6. Secondary Outcome: Anxiety Symptoms
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 8-item short form was administered. 50 indicates the population mean with a standard deviation of 10. Possible T-Scores range from 20 - 80. Higher scores indicate greater anxiety symptoms.
Time Frame: At day 14 (7 days after intervention)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
T-score | 52.91 (49.79) | 11.04 (8.84)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.49, ANOVA; Mean Difference (Final Values) = -1.02, Standard Error of Mean 1.49

7. Secondary Outcome: Depression Symptoms
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 8-item short form was administered. 50 indicates the population mean with a standard deviation of 10. Possible T-Scores range from 20 - 80. Higher scores indicate greater depression symptoms.
Time Frame: At day 7 (after intervention)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
T-score | 51.08 (9.35) | 41.31 (8.31)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.67, ANOVA; Mean Difference (Final Values) = -0.58, Standard Error of Mean 1.36

8. Secondary Outcome: Depression Symptoms
Description: as for outcome 7
Time Frame: At day 14 (7 days after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
score on a scale | 51.02 (9.36) | 48.53 (8.89)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.89, ANOVA; Mean Difference (Final Values) = -0.19, Standard Error of Mean 1.37

9. Secondary Outcome: Prescription Opioid Misuse
Description: The Current Opioid Misuse Measure (COMM), a 17-item questionnaire, was administered. Scores represent the total summed score and range from 0 to 68, with higher scores indicating greater opioid misuse
Time Frame: At day 14 (7 days after intervention)
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Coping Statement | Control
Number analyzed (Participants) | 44 | 49
total score on a scale | 8.30 (7.90) | 7.47 (6.67)
Statistical Analysis 1: Comparison: Coping Statement vs Control; Test type: Superiority; p = 0.08, ANOVA; Mean Difference (Final Values) = -1.61, Standard Error of Mean 0.90

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Coping Statement | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/49
Other Adverse Events (participants affected / at risk) | 7/44 | 13/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coping Statement (N=44) | Control (N=49)
Suicidal thought without intent (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coping Statement (N=44) | Control (N=49)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) — Includes colds/flus/throat pain
Bladder Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Pain Flare-up (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) — Includes swelling and numbness
Bodily injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Back surgery
Financial hardship (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04097743/Prot_SAP_000.pdf